CLINICAL TRIAL: NCT03042637
Title: Safety and Efficacy of Combination Acthar Gel and Tacrolimus in the Treatment of Steroid Resistant Nephrotic Syndrome
Status: Suspended | Type: Observational
Why Stopped: Bb
Sponsor: Southeast Renal Research Institute (Other)
Responsible Party: Principal Investigator, James A. Tumlin MD, Principal Investigator, Southeast Renal Research Institute
Other Study IDs: 12345
Record Dates: First submitted 2016-03-30; First posted 2017-02-03 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Tacrolimus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acthar Gel and Tacrolimus: Combination therapy with Acthar Gel and Tacrolimus
  Interventions: Drug: Acthar Gel and Tacrolimus

INTERVENTIONS:
Drug: Acthar Gel and Tacrolimus — Combination therapy with Acthar Gel and Tacrolimus (0.5-3.0 mg BID) following 6 months of ACTH therapy only

SUMMARY:
The management of steroid-resistant nephrotic syndrome (SRNS) remains a persistent problem for investigators in part because of the wide array of pathogenic cccccccccc mechanisms that contribute to these disorders as well as the lack ofs. While glucocorticoids remain the primary therapy for many forms of protein uric glomerularxxxxxxxxx diseases, prolonged use is associated with significant morbidities including steroid induced diabetes, metabolic bone disease, and excessive weight gain.

DETAILED DESCRIPTION:
Multiple agents have been investigated in the treatment of patients with SRNS, but there is no consensus on what constitutes optimal therapy. Previous studiesoids and have shown complete and partial response rates between 40% and 60%. More recently, calcineurin inhibitors (CNI) have become an effective second line therapy with similar response rates between 50%-70%. However, both treatment regiments are limited by the risk for infection as well as the development of vvvvvvv CNI-induced nephrotoxicity and progressive renal disease. Acthar gel is a porcine pituitary preparation composed of ACTH and for treatment of idiopathic nephrotic syndrome. Previous studies, as well as more current studies, have shown that ACTHar gel can effectively reduce proteinuriammmmmmmm in idiopathic membranous glomerulonephritis and other forms of glomerulopathy including focal segmental glomerulosclerosis (FSGS) and advanced diabetic nephropathy. While the mechanism is unknown, previous studies have shown that melanocortin 1-receptors are expressed in glomerular podocytes and thatpathway could be involved in the protein lowering effects of ACTHar bbbbbbbbgel. Incubation of cultured podocytes with ACTH leads to activation of MCR-1 receptors and the subsequent stimulation of protein kinase A (PKA) through a G-protein-dependent pathway. The downstream phosphorylation and stabilization of Rho GTPases, synaptopodin and other cell-cytoskeletal associated proteins may stabilize podocyte function and density.

ELIGIBILITY:
Inclusion Criteria:

* refractory nephrotic syndrome secondary, defined as subjects having a urine protein/Cr ratio over 3.0 while actively receiving ACE inhibitors and hyperglycemic therapy (i.e., insulin or oral hyperglycemic agents).
* Type I or Type II diabetes
* receiving combination therapy with an ACE inhibitor and a second protein lowering agent (e.g., ARB, non dihydropyridine CCB, or spironolactone).

Exclusion Criteria:

* known primary or secondary membranous glomerulonephritis (GN)
* primary or secondary focal segmental glomerulosclerosis
* other nondiabetic forms of glomerulopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients between the ages of 18 and 80 with refractory nephrotic syndrome secondary to Type I or Type II diabetes
Sampling Method: Non-Probability Sample
Dates: Start 2012-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of proteinuria in idiopathic membranous glomerulonephritis (MGN) and other forms of glomerulopathy including focal segmental glomerulosclerosis (FSGS) and advanced diabetic nephropathy | 6 months
  Subjects with steroid resistant nephrotic syndrome were treated with sub-cutaneous (SQ) ACTHar gel, (40-80 units) SQ 2X-3X/week. After 6 months of ACTHar gel therapy subjects achieving complete remission were weaned off therapy over a 3-12 month period.

SECONDARY OUTCOMES:
Partial remission or no response to treatment regiment | 6 months
  Subjects exhibiting no response or partial remission were maintained on existing ACTHar gel doses and started on oral Tacrolimus (0.03 to 0.06 mg/kg/day) titrating to a trough level of 5-10 ng/ml for an additional 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: James A Tumlin, MD, Principal Investigator — NephroNet Clinical Research Consortium
Locations (1):
- Nephronet, Chattanooga, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No